CLINICAL TRIAL: NCT02273609
Title: English: Current Perspective of the Status of Anticoagulation in Clinical Practice in Primare Care. Spanish: Perspectiva Actual de la sitUación de la anticoaguLación en la práctica clínica de Atención Primaria.
Brief Title: INR Control and Atrial Fibrillation in Primary Care in Spain (PAULA)
Acronym: PAULA
Status: Completed | Type: Observational
Sponsor: Vivencio Barrios (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Vivencio Barrios, MD, PhD, Hospital Universitario Ramon y Cajal
Organization: Hospital Universitario Ramon y Cajal (Other)
Other Study IDs: BAY-AVK-2013-01
Record Dates: First submitted 2014-10-18; First posted 2014-10-24 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Atrial Fibrillation and Flutter
Keywords: Atrial fibrillation; Anticoagulation; Vitamin K antagonists; INR control
MeSH Terms: conditions — Atrial Fibrillation | interventions — Acenocoumarol; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Vitamin K antagonists (acenocoumarol or warfarin) — INR values of patients treated with acenocoumarol or warfarin in the last 12 months will be recorded according to clinical practice of each center.
  No specific recommendation about treatment will be provided by sponsor.
  Other Names: acenocoumarol; warfarin

SUMMARY:
The primary objective of this study was to determine rates of INR control of patients with nonvalvular AF daily attended in primary care in Spain.

PAULA is an observational retrospective/cross-sectional and multicenter study. Patients aged ≥18 years old, with nonvalvular AF, treated with VKAs for at least one year in primary care were included in the study. To be included, at least 80% of INR values during the past 12 months should be available. Before inclusion, patients provided written consent.

Clinical data (biodemographic data, comorbidities, treatments, and thromboembolic/bleeding risk) were recorded from the clinical history of patients at the moment of inclusion. INR values were taken from the previous 12 months of inclusion.

Poor INR control was considered when percent time in therapeutic INR range (TTR) was <65% (calculated by Rosendaal method) or <60% by direct method (proportion of INR values).

A total of 1,524 patients have been included in the study.

DETAILED DESCRIPTION:
Vitamin K antagonists (VKAs) have traditionally been used for long-term prevention of thromboembolic complications in patients with atrial fibrillation (AF). Because of the variability in the dose response with VKAs and the narrow therapeutic window, monitoring the degree of anticoagulation is mandatory. The international normalized ratio (INR) provides a standardized measure of the VKA anticoagulant effect. The INR should be kept within a narrow range (therapeutic INR target 2.0-3.0) to control the intensity of anticoagulation.

The primary objective of this study was to determine rates of INR control of patients with nonvalvular AF daily attended in primary care in Spain.

PAULA is an observational retrospective/cross-sectional and multicenter study supported by the three main Spanish primary care scientific societies: Sociedad Española de Médicos de Atención Primaria (SEMERGEN), Sociedad Española de Medicina de Familia y Comunitaria (SEMFYC) and Sociedad Española de Médicos Generales y de Familia (SEMG).

Patients aged ≥18 years old, with nonvalvular AF, treated with VKAs for at least one year in primary care were included in the study. To be included, at least 80% of INR values during the past 12 months should be available. Before inclusion, patients provided written consent.

Clinical data (biodemographic data, comorbidities, treatments, and thromboembolic/bleeding risk) were recorded from the clinical history of patients at the moment of inclusion. INR values were taken from the previous 12 months of inclusion.

Poor INR control was considered when percent time in therapeutic INR range (TTR) was <65% (calculated by Rosendaal method) or <60% by direct method (proportion of INR values).

The study was approved by the ethics committee of hospital La Paz, Madrid.

A total of 1,524 patients have been included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years old with
* nonvalvular AF,
* treated with VKAs for at least one year in primary care
* At least 80% of INR values during the past 12 months should be available.
* Written consent should be provided before inclusion.

Exclusion Criteria:

* Patients that do not sign or understand written consent.
* Participating in a clinical trial in the last 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥18 years old, with nonvalvular AF, treated with VKAs for at least one year in primary care setting were included in the study.
Sampling Method: Probability Sample
Enrollment: 1524 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Anticoagulation control with vitamin K antagonists | 12 months
  international normalized ratio (INR) provides a standardized measure of the VKA anticoagulant effect. INR values of patients treated with acenocoumarol or warfarin in the last 12 months will be recorded according to clinical practice of each center.

CONTACTS AND LOCATIONS:
Overall Officials: Vivencio Barrios, MD, PhD, Principal Investigator — Hospital Ramon y Cajal

REFERENCES:
- [Result] Gallagher AM, Setakis E, Plumb JM, Clemens A, van Staa TP. Risks of stroke and mortality associated with suboptimal anticoagulation in atrial fibrillation patients. Thromb Haemost. 2011 Nov;106(5):968-77. doi: 10.1160/TH11-05-0353. Epub 2011 Sep 8. PMID 21901239
- [Result] Morgan CL, McEwan P, Tukiendorf A, Robinson PA, Clemens A, Plumb JM. Warfarin treatment in patients with atrial fibrillation: observing outcomes associated with varying levels of INR control. Thromb Res. 2009 May;124(1):37-41. doi: 10.1016/j.thromres.2008.09.016. Epub 2008 Dec 4. PMID 19062079
- [Result] Ansell J, Hollowell J, Pengo V, Martinez-Brotons F, Caro J, Drouet L. Descriptive analysis of the process and quality of oral anticoagulation management in real-life practice in patients with chronic non-valvular atrial fibrillation: the international study of anticoagulation management (ISAM). J Thromb Thrombolysis. 2007 Apr;23(2):83-91. doi: 10.1007/s11239-006-9022-7. PMID 17221328
- [Result] Clua Espuny JL, Dalmau Llorca MR, Aguilar Martin C; Grupo de Trabajo. [Characteristics of oral anti-coagulation treatment in high-risk chronic auricular fibrillation]. Aten Primaria. 2004 Nov 15;34(8):414-9. doi: 10.1016/s0212-6567(04)78925-8. Spanish. PMID 15546539
- [Result] Hess PL, Mirro MJ, Diener HC, Eikelboom JW, Al-Khatib SM, Hylek EM, Bosworth HB, Gersh BJ, Singer DE, Flaker G, Mega JL, Peterson ED, Rumsfeld JS, Steinberg BA, Kakkar AK, Califf RM, Granger CB; Atrial Fibrillation Think-Tank Participants. Addressing barriers to optimal oral anticoagulation use and persistence among patients with atrial fibrillation: Proceedings, Washington, DC, December 3-4, 2012. Am Heart J. 2014 Sep;168(3):239-247.e1. doi: 10.1016/j.ahj.2014.04.007. Epub 2014 Apr 24. PMID 25173533
- [Result] Lobos-Bejarano JM, del Castillo-Rodriguez JC, Mena-Gonzalez A, Aleman-Sanchez JJ, Cabrera de Leon A, Baron-Esquivias G, Pastor-Fuentes A; en nombre de los Investigadores del Estudio FIATE (Situacion actual de la FIbrilacion auricular en ATencion primaria en Espana). [Patients' characteristics and clinical management of atrial fibrillation in primary healthcare in Spain: FIATE Study]. Med Clin (Barc). 2013 Oct 5;141(7):279-86. doi: 10.1016/j.medcli.2012.12.023. Epub 2013 May 15. Spanish. PMID 23683967
- [Result] Melamed OC, Horowitz G, Elhayany A, Vinker S. Quality of anticoagulation control among patients with atrial fibrillation. Am J Manag Care. 2011 Mar;17(3):232-7. PMID 21504259
- [Result] Boulanger L, Kim J, Friedman M, Hauch O, Foster T, Menzin J. Patterns of use of antithrombotic therapy and quality of anticoagulation among patients with non-valvular atrial fibrillation in clinical practice. Int J Clin Pract. 2006 Mar;60(3):258-64. doi: 10.1111/j.1368-5031.2006.00790.x. PMID 16494639
- [Result] Hylek EM, Go AS, Chang Y, Jensvold NG, Henault LE, Selby JV, Singer DE. Effect of intensity of oral anticoagulation on stroke severity and mortality in atrial fibrillation. N Engl J Med. 2003 Sep 11;349(11):1019-26. doi: 10.1056/NEJMoa022913. PMID 12968085